CLINICAL TRIAL: NCT02726126
Title: Comparative Study Between Transdermal Fentanyl and Melatonin Patches on Postoperative Pain Relief After Lumber Laminectomy, a Double-blind, Placebo-controlled Trial
Brief Title: Transdermal Fentanyl and Melatonin Patches for Postoperative Pain Relief
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Dr.Ibrahim Mamdouh Esmat, Ain Shams University
Other Study IDs: 915
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Postoperative Pain
Keywords: Transdermal fentanyl; Transdermal melatonin; Postoperative pain; lumber laminectomy; Relief
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- C group, (n=25): C group, (n=25) each patient received transdermal placebo patch
  Interventions: Drug: Comparative study between transdermal fentanyl and melatonin patches on postoperative pain relief after lumber laminectomy
- TDF group, (n=25): TDF group, (n=25) each patient received transdermal therapeutic system-fentanyl 50μg/h
  Interventions: Drug: Comparative study between transdermal fentanyl and melatonin patches on postoperative pain relief after lumber laminectomy
- TDM group, (n=25): TDM group, (n=25) each patient received transdermal therapeutic system containing 7 mg of melatonin
  Interventions: Drug: Comparative study between transdermal fentanyl and melatonin patches on postoperative pain relief after lumber laminectomy

INTERVENTIONS:
Drug: Comparative study between transdermal fentanyl and melatonin patches on postoperative pain relief after lumber laminectomy

SUMMARY:
Seventy five patients, aged 18-50 years, ASA I and II undergoing elective single level lumber laminectomy under general anesthesia were included in this randomized controlled double-blind study. Patients were randomly divided into 3 groups 25 each, C group patients received transdermal placebo patch, TDF group (50μg/h) and TDM group (7 mg). Assessment of postoperative pain, sedation, hemodynamic variables such as HR and MAP, postoperative monitoring of arterial SpO2 and side effects (e.g. nausea, vomiting, pruritis, respiratory depression and hemodynamic instability) were done 30 minutes, 1, 2, 6 and 12 hours postoperatively. Postoperative Patient's and Surgeons' satisfaction, Intraoperative bleeding and plasma cortisol (µg / dl) postoperatively were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* 75 patients aged between 18 and 50 years old
* Both sex of ASA physical status I and II
* 70-90 kg body weight
* Height 160-180 cm
* Undergoing elective single level lumber laminectomy under general anesthesia.

Exclusion Criteria:

* Patients with impaired kidney or liver functions
* History of cardiac or central nervous system disease
* History of drug or alcohol abuse
* History of chronic pain or daily intake of analgesics
* Uncontrolled medical disease (diabetes mellitus and hypertension)
* History of intake of non-steroidal anti-inflammatory drugs or opioids within 24 h before surgery or allergy to the used medications
* Coagulation defect
* Local infection at the site of application of transdermal patch
* Patient refusal or duration of surgery more than 120 minutes were excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study was designed to be a randomized, placebo-controlled, double-blind parallel study in which the patients, investigators, anesthesiologists and the surgeons were blinded to the given treatment. This study was conducted in Ain-Shams university hospitals, from March 2013 to April 2015 on 75 patients aged between 18 and 50 years old of both sex of ASA physical status I and II of 70-90 kg body weight and height 160-180 cm undergoing elective single level lumber laminectomy under general anesthesia. The study protocol was approved from the institutional ethical committee and written informed consent was obtained from all the patients.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
A mean difference of total analgesic (pethidine) consumption. | The total pethidine requirements (mg) 12 hours postop